CLINICAL TRIAL: NCT03126175
Title: Above-versus Below-elbow Casting for Conservative Treatment of Distal Radius Fractures: a Randomized Controlled Trial and Study Protocol.
Brief Title: Above-versus Below-elbow Casting for Conservative Treatment of Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Dr. Fernando Mauro Pires da Rocha (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Above X below-elbow casting
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Distal Radius Fracture
Keywords: conservative treatment, treatment outcome
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Above elbow immobilization (Active Comparator): Above elbow immobililization with short radial splint that will be performed with 20cm wide gypsum cut to fit the thumb. The splint will be applied to the radial aspect of the wrist covering the volar and dorsal portion of the radius to the elbow. Additional splint with a 15cm width splint on the ulnar aspect of the forearm that begins at the middle of the forearm and extends into the armpit.
  Interventions: Device: Above elbow immobilization
- Below elbow immobilization (Experimental): Below elbow immobilization with exclusively short radial splint that will be performed with 20cm wide gypsum cut to fit the thumb. The splint will be applied to the radial aspect of the wrist covering the volar and dorsal portion of the radius to the elbow.
  Interventions: Device: Below elbow immobilization

INTERVENTIONS:
Device: Below elbow immobilization — 20cm wide gypsum in the forearm cut to fit the thumb.
  Other Names: Plaster immobilization with elbow free (Below elbow)
  Arms: Below elbow immobilization
Device: Above elbow immobilization — 20cm wide gypsum in the forearm cut to fit the thumb associated a elbow splint made with a 15cm width on the ulnar aspect of the forearm that begins at the middle of the forearm and extends into the armpit.
  Other Names: Plater immobilization including elbow (Above elbow)
  Arms: Above elbow immobilization

SUMMARY:
For the non-surgical treatment of distal radius fractures in adults a variety cast options are available, including or not the elbow joint. The literature is inconclusive regarding the need to immobilize the elbow joint after reduction of the distal radius fracture.This study was undertaken to evaluate the best method of immobilization between the above and below-elbow cast groups at the end of 6 months of follow-up.

DETAILED DESCRIPTION:
To determine the best method of immobilization ( below elbow versus above elbow splint) in patients with distal radius fractures at the end of 6 months of follow-up:

* Type of study: Prospective, randomized and controlled trial.
* Patient recruitment: Adults attended in emergency room with closed acute displaced distal radius fracture will be reduced under general venous anesthesia with fluoroscopic control.

Displaced and reducible fractures (after venous anesthesia) will be included if one of these conditions is present: Radial height - loss > 2 mm , radial Inclination- loss > 4°, dorsal tilt - > 10°, ulnar variance - loss > 3 mm, intra-articular step off or gap - > 2mm . The contralateral side will be used as a reference.

The eligible participants will be informed about the nature and purpose of the study by reading the "Informed Consent Term" after ageeement, patients will included in the trial and randomized.

* Maintenace of reduction will be defined as the maintenance of the parameters listed above.
* Patients with above elbow immobilization will remain for 4 weeks with splint followed by 2 weeks of below elbow immobilization. The immobilization will be removed with 6 weeks.
* The primary outcome is: maintenance of reduction by evaluation of radiographic parameters (wrist radiographs) at one, two, three, four, six, eight, twelve and twenty four weeks after fracture reduction and self-reported function assessment Disabilities of the Arm, Shoulder and Hand questionnaire(DASH).
* Secondary outcomes:Patient Rated Wrist Evaluation- PRWE. Pain (VAS - "Visual Analogue Pain Scale"). Objective functional evaluation (goniometry and dynamometry) and rate of complications and failures.
* Sample Size calculation was calculated based on data derived from one recent randomized clinical trial on the subject. We considered as relevant differences on DASH scores (clinically relevant) when scores are greater than 10 points and standard deviation 15 points. To detect this difference (Student T-test) and statistical power of 95% resulted in a 58 patient sample size per group. We considered an extra 10% for balancing follow up losses. Thus, our inclusion target will be 64 patients per group. We considered the test as bicaudal.

Benefits: Below elbow splinting is easier to apply, lower cost, more comfortable and permits better function for daily life activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults with growth plate closured, both gender, with closed acute displaced distal radius fracture (up to 1 week), associated or not with the ulnar styloid fractures with no other fractures, which may be closed reduced after intravenous anesthesia. No previous fractures to the ipsilateral or contralateral forearm.
* Displaced and reducible fractures (after venous anesthesia) classified by AO as type A2, A3, C1, C2 and C3.

Exclusion Criteria:

* Open fractures.
* Vascular ou neurological compromise

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
maintenance of reduction by evaluation of radiographic parameters (wrist radiographs). | One, two, three, four, six, eight, twelve and twenty four weeks after fracture reduction(radiographs).
  Posteroanterior and lateral x-rays of the wrist to measure radiographic parameters to determine maintenance of reduction will be done every follow up visit. Measurements of the alignment will be made on the radiographs with a marker, straight edge, and protractor. The radiographic measurement technique will be standardized, and repeatability testing demonstrated by a complete blinded assessor. All radiographs will be reviewed by one of the four authors.

SECONDARY OUTCOMES:
DASH questionnaire | Two, six , eight, twelve and twenty four weeks
  The DASH questionnaire was developed as an instrument for patients with upper-extremity injuries. The survey contains 37 questions related to the function of the hand, wrist, elbow, and shoulder.
Patient Rated Wrist Evaluation (PRWE) | Eight, twelve and twenty four weeks.
  The PRWE contains 15 items that are specific to determine the degree of musculoskeletal disability related to the wrist. Both are validated tools of upper extremity function.
Pain (VAS - "Visual Analogue Pain Scale"). | one, two, three, four, six, eight, twelve and twenty four weeks after fracture reduction
  Visual Analogue Pain Scale(VAS). It is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Pain in VAS is a continuous scale comprised of a horizontal line with 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]). The participants are asked to report pain intensity in the last 24 hours. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 100mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
Objective functional evaluation (goniometry and dynamometry) | Six, eight, twelve and twenty four weeks follow up visit.
  The objective functional evaluation measurement will be made with protactor to measure wrist flexion, extension, ulnar deviation, radial deviation and pronosupination

CONTACTS AND LOCATIONS:
Overall Officials: João Carlos Belloti, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Hospital Municipal Dr. Fernando Mauro Pires da Rocha, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available through contact with the researcher.
Supporting Information: Study Protocol
Time Frame: The data of study protocol is already available. doi: 10.1186/s12891-018-2007-9
Access Criteria: open
URL: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5870077/

REFERENCES:
- [Background] Bunger C, Solund K, Rasmussen P. Early results after Colles' fracture: functional bracing in supination vs dorsal plaster immobilization. Arch Orthop Trauma Surg (1978). 1984;103(4):251-6. doi: 10.1007/BF00387330. PMID 6391415
- [Background] Bong MR, Egol KA, Leibman M, Koval KJ. A comparison of immediate postreduction splinting constructs for controlling initial displacement of fractures of the distal radius: a prospective randomized study of long-arm versus short-arm splinting. J Hand Surg Am. 2006 May-Jun;31(5):766-70. doi: 10.1016/j.jhsa.2006.01.016. PMID 16713840
- [Background] Stewart HD, Innes AR, Burke FD. Functional cast-bracing for Colles' fractures. A comparison between cast-bracing and conventional plaster casts. J Bone Joint Surg Br. 1984 Nov;66(5):749-53. doi: 10.1302/0301-620X.66B5.6389558.
- [Background] Bohm ER, Bubbar V, Yong Hing K, Dzus A. Above and below-the-elbow plaster casts for distal forearm fractures in children. A randomized controlled trial. J Bone Joint Surg Am. 2006 Jan;88(1):1-8. doi: 10.2106/JBJS.E.00320. PMID 16391243
- [Background] Pool C. Colles's fracture. A prospective study of treatment. J Bone Joint Surg Br. 1973 Aug;55(3):540-4. No abstract available. PMID 4125714
- [Result] Sarmiento A, Pratt GW, Berry NC, Sinclair WF. Colles' fractures. Functional bracing in supination. J Bone Joint Surg Am. 1975 Apr;57(3):311-7. PMID 1123382
- [Derived] Okamura A, de Mendonca GM, Raduan Neto J, de Moraes VY, Faloppa F, Belloti JC. Above-versus below-elbow casting for conservative treatment of distal radius fractures: a randomized controlled trial and study protocol. BMC Musculoskelet Disord. 2018 Mar 27;19(1):92. doi: 10.1186/s12891-018-2007-9. PMID 29587687